CLINICAL TRIAL: NCT01676025
Title: Randomized Controlled Trial Between PRA(Posterior Retroperitoneoscopic Adrenalectomy) and LA(Laparoscopic Adrenalectomy)
Brief Title: Comparison Between Posterior Retroperitoneoscopic Adrenalectomy and Laparoscopic Adrenalectomy
Acronym: PRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyu Eun Lee, Assistant Professor, Department of Surgery, Seoul National University College of Medicine, Seoul, Korea, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kyu.eun.lee-001
Record Dates: First submitted 2012-08-22; First posted 2012-08-30 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Adrenal Disease
Keywords: pheochromocytoma; aldosteronism; cushing's syndrome; adrenal incidentaloma; Conn's syndrome
MeSH Terms: conditions — Adrenal Gland Diseases; Pheochromocytoma; Hyperaldosteronism; Cushing Syndrome; Adrenal incidentaloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRA (Experimental): Persons who get PRA surgery.
  Interventions: Procedure: PRA
- LA (Experimental): Persons who get LA surgery.
  Interventions: Procedure: LA

INTERVENTIONS:
Procedure: PRA
  Arms: PRA
Procedure: LA
  Arms: LA

SUMMARY:
The purpose of this study is to compare two surgical methods of adrenalectomy. One is called PRA(posterior retroperitoneal adrenalectomy), which is performed through 3 or 4 holes at patient's back. The other is LA(laparoscopic adrenalectomy) which is performed through patient's abdominal cavity after making 3 or 4 holes in the abdomen.

DETAILED DESCRIPTION:
Since 1992, transabdominal LA(laparoscopic adrenalectomy) has been a standard method of adrenalectomy. This traditional method has been used widely because this procedure provides wide view of the whole abdomen which is familiar to surgeons. But due to its unique location at retroperitoneum, adrenal is still not easy to approach. So various retroperitoneal approaches were designed and adjusted. Among those, PRA(posterior retroperitoneal adrenalectomy) has showed good outcomes in many institutes. PRA facilitates direct approach to kidney and adrenal gland, and so operative time can be shortened. But there has been no randomized controlled trial between these two methods.

Therefore, as experienced surgeons in both methods, we want to practice this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are expected to have benign adrenal disease at preoperative exams
* Patients who have pheochromocytoma measured less than 5cm, and the other benign adrenal tumors less than 7cm in diameter in preoperative CT scan
* Patients who do not have previous surgery history at the interested quadrant
* Patients who is I or II grade in ASA classification(American society of anesthesiologists' physical status classification)
* Patients who has tolerable liver function and renal function(bilirubin<2.0mg/dl and AST, ALT, serum creatinine within twice of upper normal range, coagulation panel : within normal limit)
* Patients whose BMI(body mass index) is less than 35
* Patients who are supposed to have normal cognitive function
* Patients who signed the consent paper.

Exclusion Criteria:

* Patients who are expected to have malignant or metastatic adrenal tumor at preoperative exams
* Patients who have bilateral adrenal tumors
* Patients who have condition to undergo the other operation at the abdomen together with adrenalectomy
* Pregnant patients
* Patients who have active or uncontrolled infection
* Patients who have medical problems as below
* Uncontrollable hypertension with medication(Systolic BP>150 or diastolic BP>100)
* Angina, congestive heart failure, acute myocardial infection
* History of coronary angioplasty or Coronary artery bypass graft surgery
* History of stroke, transient ischemic attack with sequela

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-09; Primary Completion 2016-02-28 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Operation time | Participants will be followed until the first visit of out patients clinic after discharge, an expected average of 3 weeks
  operation time will be measured by attending nerse

SECONDARY OUTCOMES:
Pain sensation after surgery | Participants will be followed until the first visit of out patients clinic after discharge, an expected average of 3 weeks
  Pain score will be described daily during hospitalization, and also at out patient clinic after discharge
Recovery of bowel movement | Participants will be followed the duration of hospital stay, an expected average of 5 days
  Gas out is regarded as a recovery of bowel movement
Wound complication | Participants will be followed until the first visit of out patients clinic after discharge, an expected average of 3 weeks
Blood loss during operation | Participants will be followed until the first visit of out patients clinic after discharge, an expected average of 3 weeks
Intra-operative hemodynamic status | Participants will be followed until the first visit of out patients clinic after discharge, an expected average of 3 weeks
  Events as below will be recorded and compared severe hypertension(systolic BP>200mmHg), severe hypotension(systolic BP<90mmHg), Tachycardia(HR>110/min), Bradycardia(HR<50/min)

CONTACTS AND LOCATIONS:
Overall Officials: Kyueun Lee, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Chai YJ, Yu HW, Song RY, Kim SJ, Choi JY, Lee KE. Lateral Transperitoneal Adrenalectomy Versus Posterior Retroperitoneoscopic Adrenalectomy for Benign Adrenal Gland Disease: Randomized Controlled Trial at a Single Tertiary Medical Center. Ann Surg. 2019 May;269(5):842-848. doi: 10.1097/SLA.0000000000002603. PMID 29189215